CLINICAL TRIAL: NCT02413541
Title: The Pilot Study of the Efficacy of Polymyxin-B Hemoperfusion in Critically Ill Patients With Severe Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Nattachai Srisawat ,M.D., Division of Nephrology, Department of Medicine, Faculty of Medicine, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB.575/56
Record Dates: First submitted 2015-03-31; First posted 2015-04-10 (Estimated); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Severe Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- High EAA and use Polymyxin-B Hemoperfusion (Experimental): EAA level > 0.6 or EAA = 0.6 and use Polymyxin-B Hemoperfusion
  Interventions: Procedure: Polymyxin-B Hemoperfusion
- High EAA and not use Polymyxin-B Hemoperfusion (Experimental): EAA level > 0.6 or EAA = 0.6 and not use Polymyxin-B Hemoperfusion
  Interventions: Procedure: Standard treatment
- Low EAA (Active Comparator): EAA level < 0.6 and not use Polymyxin-B Hemoperfusion
  Interventions: Procedure: Standard treatment

INTERVENTIONS:
Procedure: Polymyxin-B Hemoperfusion — Endotoxin removal
  Arms: High EAA and use Polymyxin-B Hemoperfusion
Procedure: Standard treatment
  Arms: High EAA and not use Polymyxin-B Hemoperfusion; Low EAA

SUMMARY:
This research project is a study to immunology changes in critically ill patients with severe sepsis by using Endotoxin Activity Assay (EAA) combined with Polymyxin-B Hemoperfusion.

ELIGIBILITY:
Inclusion Criteria:

* SIRS Criteria > or = 2 meets definition
* Source of infection > or = 1 meet definition
* Evidence of organ dysfunction > or = 1 meet definition

Exclusion Criteria:

* WBC < 5,000 /ul
* Platelet < 30,000 / ul
* Pregnancy woman
* Advance stage cancer patients (terminally ill) who is refuse to be resuscitated
* Received blood transfusion > 5 units in 24 hrs
* Allergy to Polymyxin-B
* High risk and uncontrolled bleeding
* Organ transplant patients
* On immunosuppressive agents within 2 weeks before study
* HIV infection

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Functions of cell surface markers | 3 days
  CD11b expression on PMN and HLA-DR expression on monocyte
Chemotaxis | 3 days
  Neutrophil function
EAA level | 3 days
  Endotoxin level

SECONDARY OUTCOMES:
Survival rate | 28 days
Sequential Organ Failure Assessment (SOFA Score) | 28 days
Acute Kidney Injury and Renal Replacement Therapy incidences | 28 days
ICU length of stay | 28 days
Mechanical ventilation free day | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Sasipha Tachaboon, Bangkok, Pathumwan, Thailand

REFERENCES:
- [Derived] Singhan W, Vadcharavivad S, Areepium N, Wittayalertpanya S, Chaijamorn W, Srisawat N. The effect of direct hemoperfusion with polymyxin B immobilized cartridge on meropenem in critically ill patients requiring renal support. J Crit Care. 2019 Jun;51:71-76. doi: 10.1016/j.jcrc.2019.02.007. Epub 2019 Feb 5. PMID 30769293
- [Derived] Srisawat N, Tungsanga S, Lumlertgul N, Komaenthammasophon C, Peerapornratana S, Thamrongsat N, Tiranathanagul K, Praditpornsilpa K, Eiam-Ong S, Tungsanga K, Kellum JA. The effect of polymyxin B hemoperfusion on modulation of human leukocyte antigen DR in severe sepsis patients. Crit Care. 2018 Oct 26;22(1):279. doi: 10.1186/s13054-018-2077-y. PMID 30367647